CLINICAL TRIAL: NCT01566526
Title: Retrospective Data Collection Study in Patients Receiving Two or More OZURDEX® Injections for Macular Oedema Secondary to Retinal Vein Occlusion
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/RET/012
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-03

CONDITIONS: Retinal Vein Occlusion; Macular Oedema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients Previously Treated with OZURDEX®: OZURDEX® administered at least twice in accordance with routine clinical practice as part of the Belgium Medical Needs Program.
  Interventions: Drug: dexamethasone intravitreal implant 0.7 mg

INTERVENTIONS:
Drug: dexamethasone intravitreal implant 0.7 mg — OZURDEX® administered at least twice in accordance with routine clinical practice as part of the Belgium Medical Needs Program.
  Other Names: OZURDEX®

SUMMARY:
The purpose of this study is to use retrospective data to evaluate the efficacy, safety and re-injection interval of OZURDEX® in the treatment of macular oedema due to retinal vein occlusion (RVO) in patients who received OZURDEX® as part of the Belgium Medical Needs Program.

ELIGIBILITY:
Inclusion Criteria:

* Macular oedema in at least one eye due to branch retinal vein occlusion (BRVO) or central retinal vein occlusion (CRVO)
* Received at least two OZURDEX® injections in the study eye as part of the Belgium Medical Needs Program

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with branch retinal vein occlusion (BRVO) or central retinal vein occlusion (CRVO) who received OZURDEX® as part of the Belgium Medical Needs Program.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Antwerp, Belgium

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Previously Treated With OZURDEX®
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Previously Treated With OZURDEX®
Number analyzed (Participants) | 26
Age, Customized [Number; unit: Participants]
  41 to 50 years | 3
  51 to 60 years | 10
  61 to 70 years | 4
  71 to 80 years | 8
  81 to 90 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to OZURDEX® Re-Injection in the Study Eye
Description: The time interval is measured from the first OZURDEX® injection to the second OZURDEX® injection in the study eye.
Time Frame: Up to 12 Months
Population: All enrolled patients.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Patients Previously Treated With OZURDEX®
Number analyzed (Participants) | 26
Days | 143.65 (42.95)

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) 7 to 12 Weeks Following Last Injection in the Study Eye
Description: BCVA is measured in the study eye following each injection of OZURDEX® using a special eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number improvement in the number of letters read means that the vision has improved. Data are reported for the 7-12 week period following the last injection.
Time Frame: Baseline, 7 to 12 weeks following the last injection
Population: All enrolled patients with data for this data point.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Patients Previously Treated With OZURDEX®
Number analyzed (Participants) | 4
Letters
  Baseline | 61.75 (29.02)
  Change from Baseline 7-12 Wks After Last Injection | -5.00 (45.28)

3. Secondary Outcome: Percentage of Patients With an Increase of 2 Lines or More in BCVA From Baseline in the Study Eye
Description: BCVA following the first injection of OZURDEX® is measured in the study eye using a special eye chart and is reported as the number of lines (5 letters per line) read correctly. An increase of 2 lines or more indicates an improvement.
Time Frame: Baseline, Up to 12 Months
Population: All enrolled patients with data for this data point.
Measure: Number; unit: Percent of Participants
Arm/Group | Patients Previously Treated With OZURDEX®
Number analyzed (Participants) | 26
Percent of Participants | 50.0

4. Secondary Outcome: Percentage of Patients With an Increase of 3 Lines or More in BCVA From Baseline in the Study Eye
Description: BCVA following the first injection of OZURDEX® is measured in the study eye using a special eye chart and is reported as the number of lines (5 letters per line) read correctly. An increase of 3 lines or more indicates an improvement.
Time Frame: Baseline, Up to 12 Months
Population: All enrolled patients with data for this data point.
Measure: Number; unit: Percent of Participants
Arm/Group | Patients Previously Treated With OZURDEX®
Number analyzed (Participants) | 26
Percent of Participants | 42.3

5. Secondary Outcome: Change From Baseline in Central Retinal Thickness in the Study Eye by Optical Coherence Tomography (OCT) 7 to 12 Weeks Following Last Injection
Description: OCT is measured in the study eye following each injection of OZURDEX®. OCT is a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina to assess retinal thickness. A negative change indicates an improvement. Data are reported for the 7-12 week period following the last injection.
Time Frame: Baseline, 7 to 12 weeks following the last injection
Population: All enrolled patients with data for this data point.
Measure: Mean (Standard Deviation); unit: Micrometers (µm)
Arm/Group | Patients Previously Treated With OZURDEX®
Number analyzed (Participants) | 6
Micrometers (µm)
  Baseline | 665.00 (287.84)
  Change from Baseline 7-12 Wks After Last Injection | -382.17 (285.36)

6. Secondary Outcome: Time to Improvement of 2 Lines or More in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: as for outcome 3
Time Frame: Baseline, Up to 12 Months
Population: All enrolled patients with data for this data point who had an improvement of ≥ 2 lines in BCVA.
Measure: Median (Full Range); unit: Days
Arm/Group | Patients Previously Treated With OZURDEX®
Number analyzed (Participants) | 13
Days | 41.0 (41.49) [25.0 to 154.0]

7. Secondary Outcome: Time to Improvement of 3 Lines or More in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: as for outcome 4
Time Frame: Baseline, Up to 12 Months
Population: All enrolled patients with data for this data point who had an improvement of ≥ 3 lines in BCVA.
Measure: Median (Full Range); unit: Days
Arm/Group | Patients Previously Treated With OZURDEX®
Number analyzed (Participants) | 11
Days | 41.0 (45.46) [25.0 to 154.0]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) related to study drug were collected from the time of the first OZURDEX® injection through six months after the last injection.
Description: All enrolled patients were used to assess adverse events (AEs) and serious adverse events (SAEs). This was a retrospective study. Patient charts were reviewed for AEs.
Arm/Group | Patients Previously Treated With OZURDEX®
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 20/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Previously Treated With OZURDEX® (N=26)
Lenticular Opacities (Eye disorders) | 5
Ocular Hypertension (Eye disorders) | 5
Intraocular Pressure Increased (Eye disorders) | 4
Cataract (Eye disorders) | 3
Cataract Operation (Eye disorders) | 3
Eye Laser Surgery (Eye disorders) | 3
Macular Fibrosis (Eye disorders) | 2
Visual Impairment (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.